CLINICAL TRIAL: NCT00029536
Title: Phase 3 Study of Progesterone vs Placebo Therapy
Brief Title: Progesterone vs Placebo Therapy for Women With Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other); Columbia University (Other); Dartmouth-Hitchcock Medical Center (Other); Emory University (Other); Johns Hopkins University (Other); Montreal Neurological Institute and Hospital (Other); Ohio State University (Other); Thomas Jefferson University (Other); University of Maryland (Other); University of Southern California (Other); University of Virginia (Other); Weill Medical College of Cornell University (Other); Minnesota Comprehensive Epilepsy Program (Unknown)
Responsible Party: Principal Investigator, Andrew Herzog, Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2001P001408; NINDS NS39466; CRC
Record Dates: First submitted 2002-01-15; First posted 2002-01-16 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Epilepsy
Keywords: Epilepsy; Seizure; Hormone; Progesterone; Catamenial
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Intervention Model Description: This was a phase III, randomized, double-blind, placebo-controlled, multicenter trial. Randomization was carried out separately for women with and without catamenial epilepsy, 2:1 to progesterone or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Catamenial Epilepsy: Progesterone Lozenges (Experimental): Subjects with catamenial epilepsy received 200 mg progesterone lozenges
  Interventions: Biological: Progesterone Lozenges
- Catamenial Epilepsy: Placebo Lozenges (Placebo Comparator): Subjects with catamenial epilepsy received matched placebo lozenges
  Interventions: Other: Matched Placebo Lozenges
- Noncatamenial Epilespy:Progesterone Lozenges (Experimental): Subjects without catamenial epilepsy received 200 mg progesterone lozenges
  Interventions: Biological: Progesterone Lozenges
- Noncatamenial Epilespy: Placebo Lozenges (Placebo Comparator): Subjects without catamenial epilepsy received matched placebo lozenges
  Interventions: Other: Matched Placebo Lozenges

INTERVENTIONS:
Biological: Progesterone Lozenges — 200mg Progesterone Lozenges
  Arms: Catamenial Epilepsy: Progesterone Lozenges; Noncatamenial Epilespy:Progesterone Lozenges
Other: Matched Placebo Lozenges — Matched Placebo Lozenges
  Arms: Catamenial Epilepsy: Placebo Lozenges; Noncatamenial Epilespy: Placebo Lozenges

SUMMARY:
The purpose of this investigation was to determine if cyclic adjunctive progesterone supplement is superior to placebo in the treatment of intractable seizures in women with and without catamenial epilepsy.

DETAILED DESCRIPTION:
This is a 6-month study. The first 3 months will gather baseline information on seizures, antiepileptic drug levels , menstrual cycles, hormone levels, emotional function, and quality of life. The second 3 months will assess the effects of treatment on these parameters.

ELIGIBILITY:
INCLUSION:

1. Subject must be between the ages of 13 and 45.
2. Subject must have a history of seizures (documented by EEG).
3. Subject must have had at least 2 seizures or auras per month during the past 3 months.
4. Subject must be on stable antiepileptic drug therapy for at least 2 months.
5. Subject must have cycle intervals between 21 and 35 days during 6 months prior to entry.

EXCLUSION:

1. Subject that is pregnant or lactating.
2. Subject that is on major tranquilizers, antidepressant medications, or reproductive hormones.
3. Subject that is unable to document seizures.
4. Subject that has progressive neurological or systemic disorder or > 2-fold elevation in liver enzyme levels

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 294 (Actual)
Dates: Start 2000-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Herzog, M.D., M.Sc., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (15):
- United States (14):
  - University of Southern California, Keck School of Medicine, Los Angeles, California
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center; Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Harvard Neuroendocrine Unit, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - MINCEP Epilepsy Care, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Presbyterian Hospital- Weill Medical College of Cornell University, Comprehensive Epilepsy Center, New York, New York
  - Columbia Medical Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson University Hospital, Comprehensive Epilepsy Center, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
- Montreal Neurological Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Herzog AG. Progesterone therapy in women with complex partial and secondary generalized seizures. Neurology. 1995 Sep;45(9):1660-2. doi: 10.1212/wnl.45.9.1660. PMID 7675223
- [Background] Herzog AG. Progesterone therapy in women with epilepsy: a 3-year follow-up. Neurology. 1999 Jun 10;52(9):1917-8. doi: 10.1212/wnl.52.9.1917-a. No abstract available. PMID 10371551
- [Background] Herzog AG, Klein P, Ransil BJ. Three patterns of catamenial epilepsy. Epilepsia. 1997 Oct;38(10):1082-8. doi: 10.1111/j.1528-1157.1997.tb01197.x. PMID 9579954
- [Result] Herzog AG, Harden CL, Liporace J, Pennell P, Schomer DL, Sperling M, Fowler K, Nikolov B, Shuman S, Newman M. Frequency of catamenial seizure exacerbation in women with localization-related epilepsy. Ann Neurol. 2004 Sep;56(3):431-4. doi: 10.1002/ana.20214. PMID 15349872
- [Derived] Maguire MJ, Nevitt SJ. Treatments for seizures in catamenial (menstrual-related) epilepsy. Cochrane Database Syst Rev. 2021 Sep 16;9(9):CD013225. doi: 10.1002/14651858.CD013225.pub3. PMID 34528245

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Catamenial Epilepsy: Progesterone Lozenges | Catamenial Epilepsy: Placebo Lozenges | Noncatamenial Epilespy:Progesterone Lozenges | Noncatamenial Epilespy: Placebo Lozenges
Started | 85 | 45 | 105 | 59
Completed | 85 | 45 | 105 | 59
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Catamenial Epilepsy: Progesterone Lozenges | Catamenial Epilepsy: Placebo Lozenges | Noncatamenial Epilespy:Progesterone Lozenges | Noncatamenial Epilespy: Placebo Lozenges | Total
Number analyzed (Participants) | 85 | 45 | 105 | 59 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (8.68) | 32.31 (8.5) | 30.71 (8.16) | 32.42 (7.87) | 31.71 (8.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 45 | 105 | 59 | 294
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent of Women Who Show a Greater Than 50% Decline in Average Daily Seizure Frequency
Description: Percent of women who show a greater than 50% decline in average daily seizure frequency
Time Frame: 9 years
Measure: Number; unit: percentage of participants
Arm/Group | Catamenial Epilepsy: Progesterone Lozenges | Catamenial Epilepsy: Placebo Lozenges | Noncatamenial Epilespy:Progesterone Lozenges | Noncatamenial Epilespy: Placebo Lozenges
Number analyzed (Participants) | 85 | 45 | 105 | 59
percentage of participants | 22.8 | 20.0 | 20.2 | 19.2

2. Secondary Outcome: Percent of Women Who Show a >50% Decline in Average Daily Seizure Frequency for the Most Severe Seizure Type.
Description: Percent of women who show a >50% decline in average daily seizure frequency for the most severe seizure type.
Time Frame: 9 years
Measure: Number; unit: percentage of participants
Arm/Group | Catamenial Epilepsy: Progesterone Lozenges | Catamenial Epilepsy: Placebo Lozenges | Noncatamenial Epilespy:Progesterone Lozenges | Noncatamenial Epilespy: Placebo Lozenges
Number analyzed (Participants) | 85 | 45 | 105 | 59
percentage of participants | 30.4 | 24.4 | 22.2 | 28.8

3. Secondary Outcome: Percentage of Women Who Show a Greater Than 50% Decline in Average Daily Seizure Frequency for Secondary Generalized, Complex Partial and Simple Partial Seizures Considered Separately
Description: Percentage of women who show a greater than 50% decline in average daily seizure frequency for secondary generalized, complex partial and simple partial seizures considered separately
Time Frame: 9 years
Measure: Number; unit: percentage of participants
Arm/Group | Catamenial Epilepsy: Progesterone Lozenges | Catamenial Epilepsy: Placebo Lozenges | Noncatamenial Epilespy:Progesterone Lozenges | Noncatamenial Epilespy: Placebo Lozenges
Number analyzed (Participants) | 85 | 45 | 105 | 59
percentage of participants
  SGMS | 39.39 | 29.41 | 21.21 | 20.83
  CPS | 23.68 | 18.60 | 21.21 | 13.73
  SPS | 41.12 | 41.21 | 42.22 | 31.82

4. Secondary Outcome: Changes in Serum Progesterone Levels in Subjects at Baseline and After Treatment.
Description: Changes in serum progesterone levels in subjects at baseline and after treatment with progesterone or placebo.
Time Frame: 9 years
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Catamenial Epilepsy: Progesterone Lozenges | Catamenial Epilepsy: Placebo Lozenges | Noncatamenial Epilespy:Progesterone Lozenges | Noncatamenial Epilespy: Placebo Lozenges
Number analyzed (Participants) | 85 | 45 | 105 | 59
ng/ml
  Baseline | 9.8 [5.8 to 12.0] | 9.1 [5.9 to 12.9] | 10.8 [7.3 to 13.1] | 9.1 [6.5 to 12.4]
  Treatment | 44.4 [28.9 to 87.9] | 9.2 [5.1 to 13.7] | 49.6 [27.0 to 88.25] | 12.0 [7.5 to 14.0]

5. Secondary Outcome: Change in Serum Levels of Antiepileptic Drugs on Progesterone and Placebo for Subjects With Catamenial and Non-catamenial Epilepsy.
Time Frame: 9 years
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Progesterone Lozenges: Subjects with catamenial and Non-Catamential epilepsy who received 200 mg progesterone lozenges
- Placebo Lozenges: Subjects with catamenial and non-Catamenial epilepsy who received matched placebo lozenges
Arm/Group | Progesterone Lozenges | Placebo Lozenges
Number analyzed (Participants) | 66 | 37
mcg/mL
  Carbamazepine | 8.9 (2.5) | 9.6 (1.8)
  Levitracetam | 23.2 (17.1) | 22.6 (12.5)
  Lamotrigine | 11.1 (8.2) | 8.4 (4.8)
  Topirimate | 10.9 (6.9) | 9.3 (4.6)
  Phenytoin | 19.7 (6.5) | 17.9 (3.9)

ADVERSE EVENTS:
Arm/Group | Catamenial Epilepsy: Progesterone Lozenges | Catamenial Epilepsy: Placebo Lozenges | Noncatamenial Epilespy:Progesterone Lozenges | Noncatamenial Epilespy: Placebo Lozenges
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/45 | 1/105 | 0/59
Serious Adverse Events (participants affected / at risk) | 3/85 | 1/45 | 3/105 | 2/59
Other Adverse Events (participants affected / at risk) | 37/85 | 23/45 | 55/105 | 27/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catamenial Epilepsy: Progesterone Lozenges (N=85) | Catamenial Epilepsy: Placebo Lozenges (N=45) | Noncatamenial Epilespy:Progesterone Lozenges (N=105) | Noncatamenial Epilespy: Placebo Lozenges (N=59)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — SUDEP
Hospitalization (General disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2) — Seizures
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catamenial Epilepsy: Progesterone Lozenges (N=85) | Catamenial Epilepsy: Placebo Lozenges (N=45) | Noncatamenial Epilespy:Progesterone Lozenges (N=105) | Noncatamenial Epilespy: Placebo Lozenges (N=59)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 3 (3) | 1 (1)
Dysepepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Nausea (General disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Vomiting (General disorders) | 2 (2) | 2 (2) | 4 (4) | 4 (4)
Fatigue (General disorders) | 14 (14) | 5 (5) | 16 (16) | 9 (9)
Nasopharyngitis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Dizziness (General disorders) | 3 (3) | 6 (6) | 7 (7) | 3 (3)
Headache (General disorders) | 3 (3) | 2 (2) | 3 (3) | 4 (4)
Depression (Psychiatric disorders) | 4 (4) | 1 (1) | 7 (7) | 2 (2)
Other (General disorders) | 5 (5) | 0 (0) | 9 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No